CLINICAL TRIAL: NCT00317837
Title: Bipolar vs. Unipolar Hemiarthroplasty for Patients Aged 70 Years or Above, With a Dislocated Medial Femoral Neck Fracture
Brief Title: Bipolar Versus Unipolar Hemiarthroplasty for Patients With a Hip Fracture
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: Recruitment was too slow, primary investigator has left the organisation
Sponsor: Northern Orthopaedic Division, Denmark (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: ON-04-005-LAM
Record Dates: First submitted 2006-04-23; First posted 2006-04-25 (Estimated); Last update posted 2014-03-31 (Estimated); Status verified 2014-03

CONDITIONS: Femoral Neck Fractures
Keywords: Fracture of Femoral Neck
MeSH Terms: conditions — Femoral Neck Fractures

ARMS (2):
- 1 (Active Comparator): Patients treated with a cemented modular hemiarthroplasty, with a unipolar head
  Interventions: Procedure: Unipolar Hemiarthroplasty of the hip joint
- 2 (Active Comparator): Patients treated with a modular cemented hemiarthroplasty with a bipolar head.
  Interventions: Procedure: bipolar hemiarthroplasty

INTERVENTIONS:
Procedure: Unipolar Hemiarthroplasty of the hip joint — Unipolar Hemiarthroplasty of the hip joint
  Arms: 1
Procedure: bipolar hemiarthroplasty — bipolar hemiarthroplasty
  Arms: 2

SUMMARY:
Insertion of a hemiarthroplasty is a well established treatment for a dislocated medial hip fracture in elderly patients. The purpose of this study is to compare unipolar and bipolar hemiarthroplasty as a treatment for patients aged 70 years or above with a dislocated medial femoral neck fracture. The study is prospective and randomised, and will be based on questionnaires, clinical examinations, registration of complications and radiographic evaluation at follow up at 3 months, 1 and 3 years postoperatively.

ELIGIBILITY:
Inclusion Criteria:

* Patients ages 70 years or above
* Dislocated medial femoral neck fracture (garden type 3-4)
* Residence in the county of Northern Jutland, Denmark

Exclusion Criteria:

* Pathologic fracture
* Failed formerly internally fixed fracture of the affected hip
* Degenerative joint disease of the affected hip or rheumatoid arthritis
* Dementia
* Terminal neoplastic disease
* No informed consent

Min Age: 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 0 (Actual)
Dates: Start 2004-10; Primary Completion 2010-12 (Estimated); Study Completion 2010-12 (Estimated)

CONTACTS AND LOCATIONS:
Overall Officials: Martin Lamm, MD, Principal Investigator — Northern Orthopaedic Division
Locations (3):
- Denmark (3):
  - Northern Orthopaedic Division, Klinik Aalborg, Aalborg, Northern Jutland
  - Northern Orthopaedic Division, Klinik Farsoe, Farsø, Northern Jutland
  - Northern Orthopaedic Division, Klinik Hjoerring, Hjørring, Northern Jutland